CLINICAL TRIAL: NCT02029755
Title: Ultrasound-guided-transversus Abdominis Plane(TAP) Block Versus Local Anesthetic(LA) Infiltration-the Effectiveness of Post-operative Pain Control in the Abdominal Surgery
Brief Title: Transversus Abdominis Plane Block Versus Local Anesthetic Infiltration for Pain Control in the Abdominal Surgery
Acronym: TAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, hsiao chien tsai, fellow researcher, Taipei Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 201309028
Record Dates: First submitted 2014-01-05; First posted 2014-01-08 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Postoperative Pain
Keywords: transversus abdominis plane block; local infiltration; ropivacaine; heart rate variability; postoperative analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Local; Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TAP block (Experimental): postoperative analgesia with sono-guided transversus abdominis plane block and intravenous patient controlled analgesia (IV-PCA). Bilateral sono-guided TAP block will be performed after the induction of general anesthesia. 20 ml of 0.25% ropivacaine will be injected to the transversus abdominis plane under ultrasound guidance at each side (total 40 ml). IV-PCA with morphine will be ready for postoperative pain control at the end of the surgery.
  Interventions: Procedure: transversus abdominis plane block; Procedure: Patient controlled analgesia
- Local infiltration (Active Comparator): postoperative analgesia with local anesthetics infiltration at surgical wound and intravenous patient controlled analgesia (IV-PCA). 20 ml of 0.5% ropivacaine will be injected at the surgical wound by the surgeon before the closure of wound. IV-PCA with morphine will be ready for postoperative pain control at the end of the surgery.
  Interventions: Procedure: local infiltration; Procedure: Patient controlled analgesia
- PCA only (Active Comparator): postoperative analgesia with intravenous patient controlled analgesia. IV-PCA with morphine will be ready for postoperative pain control at the end of the surgery.
  Interventions: Procedure: Patient controlled analgesia

INTERVENTIONS:
Procedure: transversus abdominis plane block — bilateral ultrasound-guided transversus abdominis plane block, with 20 ml of 0.25% ropivacaine at each side after the induction of general anesthesia
  Arms: TAP block
Procedure: local infiltration — local anesthetics infiltration at surgical wound with 20 ml of 0.5% ropivacaine before wound closure
  Other Names: local anesthetics infiltration
  Arms: Local infiltration
Procedure: Patient controlled analgesia — postoperative analgesia with intravenous patient controlled analgesia with morphine

SUMMARY:
Postoperative analgesia is an important part of the anesthetic care. According to the recent studies, multimodal analgesia can provide better analgesia & patient satisfaction with fewer side effect. For example, combining intravenous, intramuscular or oral analgesics with transversus abdominis plane (TAP) block or local anesthetic (LA) infiltration as the multimodal analgesia, can furnish a more effective pain control after the abdominal surgery.

For abdominal surgery, both local infiltration and TAP block target on relieving somatic pain. Local anesthetic wound infiltration is easy to perform with low risk. As the advancement of ultrasound technology, performing the TAP block also becomes easier, safer and more accurate. But whether LA infiltration or TAP block is better for the multimodal analgesia regimen remains unclear.

This study is to compare the postoperative pain score, opioid consumption, side effects, and quality of recovery between these two analgesic methods in patients undergoing abdominal surgery. The investigators hypothesized that TAP block may be more effective than LA infiltration as a part of the multimodal analgesia, and can improve the recovery after the abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult (20~65y/o)
* American Society of Anesthesiologists (ASA) physical status I~II
* Patients scheduled for regular abdominal surgery under general anesthesia

Exclusion Criteria:

* ASA physical status ≥ 3
* Allergy to morphine or local anesthetics
* Morphine tolerance
* Drug abuse or addiction
* Bleeding tendency

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chuen-Chau Chang, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan, Taiwan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAP Block | Local Infiltration | PCA Only
Started | 36 | 36 | 36
Completed | 36 | 36 | 36
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAP Block | Local Infiltration | PCA Only | Total
Number analyzed (Participants) | 36 | 36 | 36 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.17 (7.28) | 39.69 (5.38) | 42.69 (6.93) | 40.85 (6.65)
Sex/Gender, Customized [Number; unit: participants]
  Female | 36 | 36 | 36 | 108
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 36 | 36 | 36 | 108
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 36 | 36 | 36 | 108

OUTCOME MEASURES:

1. Primary Outcome: Pain Score (NRS: Numerical Rating Scale)
Description: pain scores of the participants will be followed at postoperative 1, 6, 24, 48 hour (up to 48 hours).
  (NRS: from 0 to 10, 0 = no pain, 10 = the worst pain) The higher score idicates the worse outcome.
Time Frame: postoperative 24 hour dynamic
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | TAP Block | Local Infiltration | PCA Only
Number analyzed (Participants) | 36 | 36 | 36
units on a scale | 4.50 (1.98) | 4.81 (1.77) | 4.17 (1.25)

2. Primary Outcome: Opioid Consumption
Description: opioid consumption of the participants will be followed at postoperative 1, 6, 12, 24, 36, 48 hour (up to 48 hours).
Time Frame: postoperative 48 hour
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | TAP Block | Local Infiltration | PCA Only
Number analyzed (Participants) | 36 | 36 | 36
mg | 27.69 (19.20) | 28.33 (15.89) | 21.53 (16.99)

3. Secondary Outcome: Sedation Scale
Time Frame: postoperative 1, 6, 24, 48 hour
Reporting Status: Not Posted

4. Secondary Outcome: Nausea and Vomiting Categorical Score
Time Frame: postoperative 1, 6, 24, 48 hour
Reporting Status: Not Posted

5. Secondary Outcome: Rescue Analgesic Use
Time Frame: postoperative 1, 6, 12, 24, 36, 48 hour
Reporting Status: Not Posted

6. Secondary Outcome: Rescue Antiemetics Use
Time Frame: postoperative 1, 6, 12, 24, 36, 48 hour
Reporting Status: Not Posted

7. Secondary Outcome: Time to the First Request of Analgesics
Description: participants will be followed for the duration of hospital stay
Time Frame: an expected average of 5 days
Reporting Status: Not Posted

8. Secondary Outcome: Pruritus
Time Frame: postoperative 1, 6, 24, 48 hour
Reporting Status: Not Posted

9. Secondary Outcome: Quality of Recovery 40
Time Frame: postoperative 48 hour
Reporting Status: Not Posted

10. Secondary Outcome: Heart Rate Variability
Time Frame: preoperative, postoperative 1 hour and 1 day
Reporting Status: Not Posted

11. Secondary Outcome: Time to Flatus
Description: participants will be followed for the duration of hospital stay
Time Frame: an expected average of 5 days
Reporting Status: Not Posted

12. Secondary Outcome: Length of Hospital Stay
Description: participants will be followed for the duration of hospital stay
Time Frame: an expected average of 5 days
Reporting Status: Not Posted

13. Secondary Outcome: Number of Participants With Intervention-related Complication
Description: participants will be followed for the duration of hospital stay
Time Frame: an expected average of 5 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | TAP Block | Local Infiltration | PCA Only
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No